CLINICAL TRIAL: NCT00358930
Title: A Phase 2 Study of ARQ 501 in Patients With Locally Advanced, Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study of ARQ 501 in Patients With Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 501-208
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous Cell
Keywords: squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — beta-lapachone

INTERVENTIONS:
Drug: ARQ 501

SUMMARY:
This is a Phase 2, multi-center, open label study of ARQ 501 in patients with locally advanced, recurrent or metastatic squamous cell cancer of the head and neck (SCCHN).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed and dated informed consent document prior to study-specific screening procedures.
2. Histologically or cytologically confirmed locally advanced, recurrent or metastatic SCCHN.
3. Measurable disease per RECIST.
4. ≥ 18 years old.
5. Karnofsky performance status (KPS) ≥ 70%.
6. Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last infusion of ARQ 501.
7. Hemoglobin (Hgb) ≥ 10 g/dL.
8. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (≥ 1,500/mm³).
9. Platelet count ≥ 100 x 10^9/L ( ≥ 100,000/mm³).
10. Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN) or less than or equal to 3.0 x ULN with metastatic liver disease.
11. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x ULN or less than or equal to 5.0 x ULN with metastatic liver disease.
12. Creatinine less than or equal to 1.5 x ULN.

Exclusion Criteria:

1. Primary tumor of nasopharyngeal origin.
2. Eligible for curative surgery or radiotherapy.
3. Received three or more systemic anticancer regimens.
4. Have active, uncontrolled systemic infection considered opportunistic, life threatening or clinically significant at the time of treatment.
5. Have received anticancer chemotherapy, immunotherapy, radiotherapy, or investigational agents within three weeks of first infusion.
6. Surgery within two weeks of first infusion.
7. Have symptomatic or untreated central nervous system (CNS) involvement.
8. Are pregnant or lactating.
9. Previous exposure to ARQ 501.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Assess the overall response rate (ORR) of patients with locally advanced, recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) treated with ARQ 501.

SECONDARY OUTCOMES:
Determine the progression-free survival (PFS) at six months for those patients treated with ARQ 501.To further characterize the safety ARQ 501.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of South Alabama, Mobile, Alabama
  - LA County Hospital, Los Angeles, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - New York Oncology Hematology, Albany, New York
  - Mary Crowley Medical Research Center, Dallas, Texas